CLINICAL TRIAL: NCT05194748
Title: Correlation of Diaphragmatic Thickness With Pulmonary Function in Parkinson's Disease
Brief Title: Diaphragmatic Thickness and Pulmonary Function in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ramazan KURUL, Assistant Professor, Abant Izzet Baysal University
Other Study IDs: AIBU-FTR-ETB-002
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Parkinson's Disease and Parkinsonism
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- camptocormia group: Diaphragmatic thickness will be measured by ultrasonography. Respiratory function will be evaluated by spirometric measurements. Postural deviations of the spine, knees, and hips will be recorded through photographs taken from the side and back
  Interventions: Other: No intervention, observational only
- no camptocormia group: Diaphragmatic thickness will be measured by ultrasonography. Respiratory function will be evaluated by spirometric measurements. Postural deviations of the spine, knees, and hips will be recorded through photographs taken from the side and back
  Interventions: Other: No intervention, observational only

INTERVENTIONS:
Other: No intervention, observational only — No intervention, observational only

SUMMARY:
Ultrasound can give important information about the morphology of the diaphragm and the amount of contraction. Our aim, with the prediction that a restrictive pathology will occur in the pulmonary function with the addition of camptocormia in Parkinson's patients; to compare respiratory functions in Parkinson's patients with and without camptocormia, to investigate the correlation between ultrasonographically measured diaphragmatic thickness and pulmonary function test values.

DETAILED DESCRIPTION:
Respiratory complications are one of the most common causes of death in Parkinson's patients. In Parkinson's disease, abnormal flexion of the thoracolumbar spine of 45° or more, which is called camptocormia, increases during walking or standing and disappears completely in the supine position. The prevalence of camptocormia among Parkinson's patients is about 7%. Camptocormia in Parkinson's disease is associated with significant disease disability, higher daily dopaminergic drug dosage, and cognitive impairment. Parkinson's patients with camptocormia often complain of shortness of breath, attributed to reduced pulmonary capacity due to limited chest expansion. Diaphragmatic dyskinesia in Parkinson's patients may also lead to a restrictive deterioration in respiratory functions.

Diaphragmatic thickness indicates diaphragmatic contraction and is correlated with PFT. Our aim; It is a comparison of respiratory functions in Parkinson's patients with and without camptocormia.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Parkinson's
* Volunteer to participate in the study

Exclusion Criteria:

* Being in contact with or suffering from COVID-19
* Having diseases that increase intra-abdominal pressure and venous insufficiency
* Having diseases that affect diaphragmatic motility
* Have had recent thoracic or abdominal surgery
* Having a parenchymal, pleural, or chest wall mass that may cause restriction on a recent chest X-ray or CT

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with Parkinson's Disease in our clinic between June 2021 and January 2023.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2021-12-24 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Pulmonary function test | 1 hour
  When the patient is in the suIt will be evaluated by conventional spirometric measurements. Pulmonary function tests will be applied to all individuals in a sitting position with the "Vmax Encore PFT system, Carefusion, CA USA" brand test device. In each measurement, the maneuvers will be repeated at least 3 times and the best values will be recorded. Forced vital capacity (FVC), expire in the first second of forced expiration (FEV1), and the ratio of FEV1 to FVC (FEV1/FVC) will be recorded.pine position, by placing a transducer on the chest wall at the level of the right 9th intercostal space, diaphragmatic movement will be monitored during inspiration, and diaphragmatic thickness will be measured at the end of expiration and inspiration. Thrombus location was evaluated proximal and/or distally by performing Doppler ultrasound
Ultrasonography | 1 hour
  When the patient is in the supine position, by placing a transducer on the chest wall at the level of the right 9th intercostal space, diaphragmatic movement will be monitored during inspiration, and diaphragmatic thickness will be measured at the end of expiration and inspiration. Thrombus location was evaluated proximal and/or distally by performing Doppler ultrasound

SECONDARY OUTCOMES:
Camptocormia measurement | 1 hour
  Postural deviations of the spine, knees and hips will be recorded through photographs taken from the side and back in the standing position. The individual's flexion of more than 45° from the thoracolumbar spine will be recorded as the presence of camptocormia. Waist, right and left knee circumference measurements also recorded

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Kurul, Ph.D, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Abant Izzet Baysal University Faculty of Health Science, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No